CLINICAL TRIAL: NCT00069758
Title: A Multi-Center Phase II Study to Investigate the Safety and Activity of SDX-105 (Bendamustine) in Patients With Indolent Non-Hodgkin's Lymphoma (NHL) Who Are Refractory to Rituximab
Brief Title: Safety and Activity of SDX-105 (Bendamustine) in Patients With Rituximab Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDX-105-01; NCT00085033 (obsolete NCT alias)
Record Dates: First submitted 2003-09-30; First posted 2003-10-02 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NHL, indolent NHL, non-Hodgkin's lymphoma, lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Bendamustine Hydrochloride

INTERVENTIONS:
Drug: SDX-105

SUMMARY:
Summary: As this is an open label study, all patients will receive SDX-105 by 30-60 minute intravenous infusion on day 1 and day 2. Treatment will repeat every 21 days. Treatment can continue for up to one year in the absence of disease progression or unacceptable toxicity. Patients will be followed until disease progression.

Rationale: Drugs used in chemotherapy, such as SDX-105, use different ways to stop tumor cells from dividing so they stop growing or die.

Purpose: This study will evaluate the effectiveness and safety in non-Hodgkin's lymphoma in patients who are refractory to Rituxan.

ELIGIBILITY:
Inclusion Criteria:

* Documented indolent or transformed B-Cell NHL indolent NHL: follicular B-Cell lymphoma, diffuse small lymphocytic lymphoma, lymphoplasmacytic lymphoma, marginal zone lymphoma
* Documented refractory disease to rituximab therapy, given as a single agent or in combination (defined as no response, or progression within 6 months of completing rituximab treatment.)
* Age of at least 18 years at Screening Visit (Site specific requirement may differ)

Exclusion Criteria:

* Previous chemotherapy or immunotherapy within 3 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin) or failure to recover from adverse events due to any agents administered previously.
* Use of investigational agents within 28 days of study
* History of prior high dose chemotherapy with allogeneic stem cell support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2003-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Comprehensive Cancer Center-Desert Regional Medical Center, Palm Springs, California
  - San Diego Cancer Center, Vista, California
  - Georgetown University Medical Center - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Mountain States Tumor Institute, Boise, Idaho
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
- Canada (4):
  - Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - CHA Hopital Enfant-Jesus, Québec, Quebec